CLINICAL TRIAL: NCT02584868
Title: Colloids in Pediatric Cardiac Surgery: Comparison Between a Balanced and a Non-balanced Colloid
Acronym: COLCHIRCARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-006034-17
Record Dates: First submitted 2013-07-03; First posted 2015-10-23 (Estimated); Results first posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2017-02

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; Sodium Chloride; HES 130-0.4

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volulyte (Experimental): Investigational drug: HES 130/0.4 (6%) in an isotonic electrolyte solution (brand name=Volulyte®)
  Interventions: Drug: Hydroxyethyl starch 130/0.4 in an isotonic electrolyte solution
- Voluven (Active Comparator): Control drug: HES 130/0.4 (6%) in sodium chloride 0.9% (brand name=Voluven®)
  Interventions: Drug: Hydroxyethyl starch 130/0.4 in 0.9% sodium chloride

INTERVENTIONS:
Drug: Hydroxyethyl starch 130/0.4 in an isotonic electrolyte solution — Peri-operative fluid replacement therapy (max 40ml/kg/day)
  Other Names: Volulyte
  Arms: Volulyte
Drug: Hydroxyethyl starch 130/0.4 in 0.9% sodium chloride — Peri-operative fluid replacement therapy (max 40ml/kg/day)
  Other Names: Voluven
  Arms: Voluven

SUMMARY:
This study will compare the clinical efficacy and safety of Volulyte® and Voluven® during elective open-heart surgery in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 28 days to 3 years old
* Planned cardiac surgery with cardiopulmonary by-pass
* signed informed consent

Exclusion Criteria:

* Moribund patients (ASA 5)
* Jehovah Witnesses
* Pre-operative coagulation disorders
* Pre-operative renal insufficiency
* Pre-operative hepatic disorders
* Intra-cranial hemorrhage
* hypernatremia

Ages: 28 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2013-02-15 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2016-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van der Linden, MDPhD, Principal Investigator — HUDERF
Locations (1):
- Hôpital Universitaire Des Enfants Reine Fabiola, Brussels, Belgium

REFERENCES:
- [Derived] Willems A, De Groote F, Schmartz D, Fils JF, Van der Linden P. Does a balanced colloid decrease perioperative blood loss in paediatric cardiac surgery: A double-blinded randomized controlled trial? Eur J Anaesthesiol. 2021 Sep 1;38(9):923-931. doi: 10.1097/EJA.0000000000001526. PMID 33966019

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline Colloid: 6% Hydroxyethyl starch 130/0.4 in NaCl 0.9% (Voluven®)
- Balanced Colloid: 6% hydroxyethyl starch 130/0.4 in an isotonic solution of electrolytes (Volulyte®)
Period: Overall Study
Arm/Group | Saline Colloid | Balanced Colloid
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Children undergoing cardiac surgery with cardiopulmonary bypass - perioperative period
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Colloid | Balanced Colloid | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 44 | 88
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 6.3 [4.5 to 13.7] | 6.9 [5.2 to 16.1] | 6.6 [5.0 to 15.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 20 | 26 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: Calculated Blood Loss at 3rd Post Operative Day (POD)
Time Frame: 72H post surgery
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
ml/kg | 19.9 [13.8 to 26.1] | 15.9 [9.0 to 25.3]

2. Secondary Outcome: Intraoperative Blood Loss
Description: peri-operative blood losses in ml/kg at the end of surgery
Time Frame: End of surgery, an average of 200 minutes
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
ml/kg | 4.7 [2.8 to 7.2] | 4.8 [2.9 to 6.4]

3. Secondary Outcome: Chest Tube Drainage
Description: Total chest tube drainage during Pediatric Intensive Care Unit (PICU) stay
Time Frame: 72H post surgery
Measure: Mean (Inter-Quartile Range); unit: ml/kg
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
ml/kg | 18.8 [11.8 to 27.7] | 18.8 [14.8 to 28.3]

4. Secondary Outcome: Total Blood Loss
Description: Total blood loss Intraoperative + chest tube drainage during Pediatric Intensive Care Unit (PICU) stay
Time Frame: 72H post surgery
Measure: Mean (Inter-Quartile Range); unit: ml/kg
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
ml/kg | 25.7 [18.7 to 34.0] | 23.4 [18.4 to 34.1]

5. Secondary Outcome: Exposure to Any Blood Products
Description: Transfusion of any blood product (intraoperative + during Pediatric Intensive Care Unit stay)
Time Frame: 72H post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
Participants | 36 | 30

6. Secondary Outcome: Exposure to Red Blood Cell
Description: Transfusion of Red Blood Cell (intraoperative + during Pediatric Intensive Care Unit stay)
Time Frame: 72H post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
Participants | 35 | 30

7. Secondary Outcome: Red Blood Cell Transfused
Description: Red Blood Cell transfused in transfused patients in ml/kg (intraoperative + during Pediatric Intensive Care Unit stay)
Time Frame: 72H post surgery
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 35 | 30
ml/kg | 21.9 [18.4 to 38.5] | 26.1 [15.7 to 44.4]

8. Secondary Outcome: Exposure to Fresh Frozen Plasma
Description: Transfusion of Fresh Frozen Plasma (intraoperative and during Pediatric Intensive Care Unit stay)
Time Frame: 72H post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
Participants | 4 | 4

9. Secondary Outcome: Fresh Frozen Plasma Transfused
Description: Fresh Frozen Plasma transfusion in ml/kg (intraoperative and during Pediatric Intensive Care Unit stay)
Time Frame: 72H post surgery
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 4 | 4
ml/kg | 12.6 [9.3 to 46.4] | 12.2 [10.1 to 26.8]

10. Secondary Outcome: Exposure to Platelets
Description: Transfusion of platelets (intraoperative and during Pediatric Intensive Care Unit stay)
Time Frame: 72H post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
Participants | 2 | 0

11. Secondary Outcome: Platelet Transfused
Description: Platelet transfusion in ml/kg (intraoperative and during Pediatric Intensive Care Unit stay)
Time Frame: 72H post surgery
Population: No platelet transfusion performed in subjects enrolled in the balanced colloid group
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 2 | 0
ml/kg | 13.7 (6.4) |

12. Secondary Outcome: Creatinine
Time Frame: At admission to the pediatric intensive care unit (Hour 0 Day 0 after surgery)
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 0.28 [0.24 to 0.33] | 0.29 [0.25 to 0.36]

13. Secondary Outcome: C-Reactive Protein (CRP)
Time Frame: At admission to the pediatric intensive care unit (Hour 0 Day 0 after surgery)
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 5.0 [1.4 to 5.0] | 5.0 [1.8 to 5.0]

14. Secondary Outcome: PTT
Time Frame: End of surgery, an average of 200 minutes
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
percent | 52.1 (9.4) | 50.1 (10.4)

15. Secondary Outcome: APTT
Time Frame: End of surgery, an average of 200 minutes
Measure: Mean (Standard Deviation); unit: seconde
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
seconde | 39.4 (5.8) | 38.6 (5.0)

16. Secondary Outcome: INR
Time Frame: End of surgery, an average of 200 minutes
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
ratio | 1.5 [1.4 to 1.7] | 1.5 [1.4 to 1.7]

17. Secondary Outcome: Fibrinogen
Time Frame: End of surgery, an average of 200 minutes
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 159.0 (51.0) | 148.0 (38.0)

18. Secondary Outcome: Clotting Time in Seconds
Description: Clotting time on EXTEM ROTEM®
Time Frame: End of surgery, an average of 200 minutes
Measure: Median (Inter-Quartile Range); unit: secondes
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
secondes | 90.5 [72.8 to 111.3] | 88.0 [59.0 to 103.5]

19. Secondary Outcome: Maximal Cloth Firmness
Description: Maximal cloth firmness on EXTEM ROTEM®
Time Frame: End of surgery, an average of 200 minutes
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mm | 50.0 [42.8 to 55.0] | 48.0 [42.0 to 52.5]

20. Secondary Outcome: Creatinine
Time Frame: Post-operative Day 1
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 0.33 [0.24 to 0.46] | 0.30 [0.26 to 0.42]

21. Secondary Outcome: CRP
Time Frame: Post-operative Day 1
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 31.3 [23.5 to 45.0] | 39.5 [25.8 to 56.0]

22. Secondary Outcome: PTT
Time Frame: Post-operative Day 1
Measure: Mean (Inter-Quartile Range); unit: percent
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
percent | 87.5 [75.0 to 96.8] | 81.0 [71.0 to 99.0]

23. Secondary Outcome: APTT
Time Frame: Post-operative Day 1
Measure: Mean (Inter-Quartile Range); unit: seconde
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
seconde | 31.2 [28.9 to 35.7] | 34.7 [31.1 to 38.9]

24. Secondary Outcome: INR
Time Frame: Post-operative Day 1
Measure: Mean (Inter-Quartile Range); unit: ratio
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
ratio | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.2]

25. Secondary Outcome: Fibrinogen
Time Frame: Post-operative Day 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 345.0 (83.0) | 365.0 (94.0)

26. Secondary Outcome: Creatinine
Time Frame: Post-operative Day 2
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 0.29 [0.22 to 0.34] | 0.27 [0.22 to 0.33]

27. Secondary Outcome: CRP
Time Frame: Post-operative Day 2
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 41.0 [23.2 to 55.6] | 43.5 [27.4 to 65.3]

28. Secondary Outcome: PTT
Time Frame: Post-operative Day 2
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
percent | 86.0 [72.0 to 96.0] | 80.5 [71.8 to 97.5]

29. Secondary Outcome: APTT
Time Frame: Post-operative Day 2
Measure: Median (Inter-Quartile Range); unit: seconde
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
seconde | 31.5 [28.7 to 35.7] | 33.2 [29.2 to 36.7]

30. Secondary Outcome: INR
Time Frame: Post-operative Day 2
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
ratio | 1.1 [1.0 to 1.2] | 1.1 [1.0 to 1.2]

31. Secondary Outcome: Fibrinogen
Time Frame: Post-operative Day 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 346.2 (82.2) | 352.6 (90.5)

32. Secondary Outcome: Creatinine
Time Frame: Post-operative Day 3
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 0.25 [0.18 to 0.32] | 0.24 [0.19 to 0.29]

33. Secondary Outcome: CRP
Time Frame: Post-operative Day 3
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Saline Colloid | Balanced Colloid
Number analyzed (Participants) | 44 | 44
mg/dl | 33.0 [22.0 to 53.7] | 29.6 [19.8 to 49.5]

ADVERSE EVENTS:
Time Frame: through study completion, an average of 14 days
Arm/Group | Saline Colloid | Balanced Colloid
All-Cause Mortality (participants affected / at risk) | 1/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/44
Other Adverse Events (participants affected / at risk) | 14/44 | 10/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saline Colloid (N=44) | Balanced Colloid (N=44)
Heart Failure (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saline Colloid (N=44) | Balanced Colloid (N=44)
Renal failure (Renal and urinary disorders) | 2 | 3
Convulsion (Nervous system disorders) | 0 | 2
Hyponatremia (Na<130) (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Na>150) (Metabolism and nutrition disorders) | 1 | 3
Hyperchloremia (Cl>115) (Metabolism and nutrition disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes